CLINICAL TRIAL: NCT04500925
Title: The Incidence of Postoperative Re-stratification for Recurrence in Well-differentiated Thyroid Cancer - A Single Tertiary Israeli Center Experience
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-20-NC-TLV-704-16-CTIL
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Well Differentiated Thyroid Carcinoma; Papillary Thyroid Cancer
Keywords: Low risk, Risk stratification, Partial thyroidectomy, Hemithyroidectomy, Completion Thyroidectomy
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UPSCALED
  Interventions: Procedure: UNILATERAL THYROIDECTOMY
- NOT UPSCALED
  Interventions: Procedure: UNILATERAL THYROIDECTOMY

INTERVENTIONS:
Procedure: UNILATERAL THYROIDECTOMY
  Other Names: TOTAL THYROIDECTOMY

SUMMARY:
Background After diagnosing well-differentiated thyroid cancer (WDTC), careful assessment of the risk for disease-specific recurrence is essential for deciding between partial (low risk) and completion (high risk) thyroidectomies. Patients' preoperatively determined risk levels are re-stratified according to surgical and final histopathological findings. The American Thyroid Association 2015 guidelines suggest that patients with WDTC between 1-4 cm in size and without suspicious features may be suitable candidates for partial thyroidectomy. The incidence and clinical implications of high-risk features discovered postoperatively in patients with preoperatively determined low-risk WDTC have not been previously reported.

Methods All thyroidectomies performed between 2006-2018 in the Tel Aviv Sourasky Medical Center were included. Pre- and postoperative risk stratifications were performed, and the rate of completion thyroidectomy was determined. Patients with 1-4 cm WDTC without evidence of positive cervical lymph nodes, invasion to adjacent structures, or high-risk cytology were considered at low risk for disease-specific recurrence and therefore suitable for lobectomy.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent thyroid surgery (partial and total) between 2006-2018 at Tel Aviv Sourasky Medical Center (TASMC) were included

Exclusion Criteria:

* Patients with evidence of cervical lymph node metastasis, other malignancies, adverse imaging features (i.e., extracapsular spread of thyroid malignancy, vocal cord paralysis or immobility in physical examination) were excluded from the study.

Ages: 38 Years to 61 Years | Sex: All
Age Groups: Adult
Study Population: The medical charts of all patients who underwent thyroid surgery between January 2006 and December 2018 in TASMC were retrieved. Most of them were females. The mean age of the entire cohort was 49.59 ± 15.17 years (median 50 years, interquartile range 38-61].
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
disease-specific recurrence | 2006-2018
  WDTC recurrence